CLINICAL TRIAL: NCT04723485
Title: Evaluation Study: Obsessive-compulsive Disorders in Childhood and Young Adulthood
Status: Recruiting | Type: Observational
Sponsor: Susanne Walitza (Other)
Responsible Party: Sponsor-Investigator, Susanne Walitza, Head of the Department of Child and Adolescent Psychiatry, Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Other Study IDs: KJPP 2019-00230
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obsessive-compulsive disorders are very damaging illnesses that can already manifest in childhood and adolescence. With an average prevalence from 1 - 3%, they are one of the most frequently diagnosed psychiatric illness in these age groups. With the further use of data, the treatment success can be significantly improved; causal variables/predictors can be recognized, understood and taken carefully into account. The anticipated incremental knowledge will ultimately help children and young people with obsessive-compulsive disorders to receive faster and more effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children and young people from 8-18 years of age who fulfill the international classification of diseases tenth edition (ICD-10) , obsessive-compulsive disorder handled in our clinic.
* Good German language speaking skills
* IQ > 75
* All study participants or their legal representative have given written permission for their experiences to be documented in the study.

Exclusion Criteria:

* Schizophrenia-related disorders (psychoses)
* Missing data
* Data sets without confirmed diagnosis
* Purely consultaive patient interview (no therapy intervention prescribed)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The sample consist of pupils with obsessive-compulsive disorder 4 to 18 years
Sampling Method: Non-Probability Sample
Enrollment: 625 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Symptoms severity of obsessive and compulsive symptoms in children and adolescents | 24 months
  The clinician report questionnaire (BY-BOCS) contains 19 items designed to assess severity of obsessive and compulsive symptoms in children and adolescents.The test uses a four point scale to rate the severity of their obsessive compulsive behaviors. Higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Walitza, Prof. Dr. med. Dipl.-Psych., Principal Investigator — Sponsor-Investigator
Locations (1):
- Psychiatric University Clinics, Department of Child and Adolescent Psychiatry, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided